CLINICAL TRIAL: NCT05748652
Title: Clinical Effectiveness of Digital CBT for the Treatment of Generalized Anxiety Disorder: A Randomized Controlled Trial
Brief Title: Generalized Anxiety Therapy Effectiveness
Acronym: GATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Big Health Inc. (Industry)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BH-D-01
Record Dates: First submitted 2023-02-17; First posted 2023-03-01 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-12

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; GAD; anxiety; digital CBT
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Digital CBT (Experimental): digitally-delivered CBT for anxiety accessed via mobile app
  Interventions: Device: digital CBT
- Psychoeducation (Active Comparator): psychoeducation delivered via digital written materials
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Device: digital CBT — An app-based intervention based on principles from cognitive behavioral therapy for anxiety.
  Arms: Digital CBT
Other: Psychoeducation — Participants will be provided with psychoeducation which will be delivered digitally upon allocation to the psychoeducation arm.
  Arms: Psychoeducation

SUMMARY:
This study will examine the effectiveness of digital CBT versus psychoeducation in improving anxiety for those with Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
This study aims to examine the effectiveness of app-based digital CBT for anxiety compared to psychoeducation in individuals with a diagnosis of Generalized Anxiety Disorder. The primary outcomes are anxiety symptom reduction and remission after 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥22 years old
* Score ≥15 on the 7-item Generalized Anxiety Disorder questionnaire (GAD-7)
* Diagnosis of GAD
* Current resident of the USA
* Oral and written fluency in English
* Regular access to the internet via a mobile or tablet device using Android ( 8 or higher) or iOS (13 or higher)
* Participant is able and willing to comply with protocol requirements, has been informed of the nature of the study, and has signed the IRB-approved informed consent form

Exclusion Criteria:

* Must not be currently receiving or be expecting to start psychological treatment for anxiety during study participation, or have previously received Cognitive Behavioral Therapy (CBT) or Acceptance and Commitment Therapy (ACT) for anxiety in the past 6-months (self-report)
* If on psychotropic medication, this must be stable for at least 60 days
* Past or present psychosis, schizophrenia, or bipolar disorder, or current OCD
* Past 12 months alcohol or substance use disorder of moderate or greater severity
* Moderate or greater suicide risk
* Hearing or vision impairment that prevents effective use of the audio-visual content of digital CBT or psychoeducation
* Intellectual disability or any Neurocognitive or Neurodevelopmental disorder that would prevent participants from following study procedures
* Any condition that the investigator believes would make participation in the study not in the best interest of the subject or would preclude successful completion of study activities

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder Questionnaire (GAD-7) | 10 weeks post-randomization
  Validated questionnaire; a 7-item scale with total scores between 0 and 21 where higher scores indicate greater severity
Generalized Anxiety Disorder remission (score 1 or 2) on the the Clinical Global Impression Scale - Improvement (CGI-I) | 10 weeks post-randomization
  A single-item measure scored between 1 and 7 where scores of 1 or 2 indicates clinically significant improvement, a score of 3 indicates mild improvement, a score of 4 indicates no change, and scores from 5 to 7 indicate deterioration

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Questionnaire (GAD-7) | 6 and 24 weeks post-randomization
  Validated questionnaire; a 7-item scale with total scores between 0 and 21 where higher scores indicate greater severity
Generalized Anxiety Disorder remission (score 1 or 2) on the the Clinical Global Impression Scale - Improvement (CGI-I) | 24 weeks post-randomization
  A single-item measure scored between 1 and 7 where scores of 1 or 2 indicates clinically significant improvement, a score of 3 indicates mild improvement, a score of 4 indicates no change, and scores from 5 to 7 indicate deterioration
Patient Health Questionnaire (PHQ-8) | Weeks 10 and 24 post-randomization
  Validated questionnaire; an 8-item scale with total scores between 0 and 24 where higher scores indicate greater severity
Sleep Condition Indicator (SCI-8) | Weeks 10 and 24 post-randomization
  Validated questionnaire; an 8-item scale with total scores between 0 and 32 where higher scores indicate better sleep
Clinical Global Impression - Severity (CGI-S) | Weeks 10 and 24 post-randomization
  A single-item measure scored between 1 and 7 where higher scores indicate greater severity of Generalized Anxiety Disorder Symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parsons EM, Ball T, Carl J, Henry AL, Emsley R, Miller CB, Wong EY, Coombs E, Collins D, Long LJ, Ster AC, Smits JAJ, Otto MW. Digital Cognitive Behavioral Treatment for Generalized Anxiety Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2548884. doi: 10.1001/jamanetworkopen.2025.48884. PMID 41396602